CLINICAL TRIAL: NCT00102284
Title: Improved Language Acquisition Through Neuromodulation, Project Stage Ia
Brief Title: Neuromodulation and Language Acquisition (Project Stage Ia)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS-NEUROMOD_01, Stage Ia; IZKF Muenster: Kne3/074/04
Record Dates: First submitted 2005-01-26; First posted 2005-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2006-09

CONDITIONS: Healthy
Keywords: language acquisition; plasticity; stroke recovery; associative learning
MeSH Terms: interventions — Levodopa; Rivastigmine; Modafinil

INTERVENTIONS:
Drug: levodopa
Drug: rivastigmine
Drug: pergolid
Drug: modafinil

SUMMARY:
The purpose of this study is to determine whether levodopa, pergolid, rivastigmine, or modafinil are effective in boosting semantic language acquisition in healthy subjects.

DETAILED DESCRIPTION:
Our prior work shows that d-amphetamine and the dopamine precursor levodopa markedly improve word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind clinical trial, we probe whether a mixed d1/d2 dopamine agonist (pergolid) or cholinergic neuromodulation (rivastigmine) or a general centrally arousing substance (modafinil) will yield a learning enhancement comparable to using levodopa in healthy subjects.

Our results show that the dopamine agonist pergolide impaired learning in healthy subjects compared to placebo, whereas cholinergic neuromodulation had no effect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* 20-35 years old
* Right handedness
* Left language dominance (as assessed by functional transcranial Doppler ultrasonography [fTCD])

Exclusion Criteria:

* Neurological/psychiatric/metabolic/cardiac disorders
* Asthma
* Known allergic reactions to one of the experimental drugs
* Other drugs affecting the central nervous system
* Leisure drug ingestion during the past 4 weeks (urine test)
* Smoking cessation during the past 2 weeks
* > 6 cups of coffee or energy drinks per day
* > 10 cigarettes per day
* > 50 grams of alcohol per day

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2005-04

PRIMARY OUTCOMES:
Boost in language learning success through neuromodulation

SECONDARY OUTCOMES:
Stability of language learning success

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Breitenstein, PhD, Study Director — Dept. of Neurology, University Hospital Muenster; Stefan Knecht, MD, Study Chair — Dept. of Neurology, University Hospital Muenster
Locations (1):
- Dept. of Neurology, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Wailke S, Bushuven S, Kamping S, Zwitserlood P, Ringelstein EB, Knecht S. D-amphetamine boosts language learning independent of its cardiovascular and motor arousing effects. Neuropsychopharmacology. 2004 Sep;29(9):1704-14. doi: 10.1038/sj.npp.1300464. PMID 15114342
- [Background] Breitenstein C, Floel A, Korsukewitz C, Wailke S, Bushuven S, Knecht S. A shift of paradigm: from noradrenergic to dopaminergic modulation of learning? J Neurol Sci. 2006 Oct 25;248(1-2):42-7. doi: 10.1016/j.jns.2006.05.012. Epub 2006 Jul 11. PMID 16815467
- [Background] Korsukewitz C, Breitenstein C, Schomacher M, Knecht S. [Present status and future possibilities of adjuvant pharmacotherapy for aphasia]. Nervenarzt. 2006 Apr;77(4):403-15. doi: 10.1007/s00115-005-2006-6. German. PMID 16273340
- [Result] Breitenstein C, Korsukewitz C, Floel A, Kretzschmar T, Diederich K, Knecht S. Tonic dopaminergic stimulation impairs associative learning in healthy subjects. Neuropsychopharmacology. 2006 Nov;31(11):2552-64. doi: 10.1038/sj.npp.1301167. Epub 2006 Jul 26. PMID 16880771